CLINICAL TRIAL: NCT05419752
Title: Assessment of 3 Different Root Canal Obturating Sealers on Postoperative Pain and Swelling in Single Canal Necrotic Teeth With a Single Visit .a Randomized Controlled Trial
Brief Title: Clinical Assessment of 3 Differant Obturation Sealers on Postoprative Pain and Swelling
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Elsayed Hany Elsayed Attia Elmasry, Master's degree student - faculty of dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENDO 23/5/2022
Record Dates: First submitted 2022-05-27; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Necrotic Pulp; Single Root Teeth
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — EndoSequence root repair material; Pemetrexed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- endo sequence bioceramic sealer (Experimental): obturation using Endo-sequence BC sealer
  Interventions: Drug: bioceramic sealer
- MTA fill apex calcium silicate base sealer (Experimental): obturation using calcium-silicates based MTA fill-apex sealer
  Interventions: Drug: MTA
- AH plus resin sealer (Experimental): obturation using AH Plus sealer
  Interventions: Drug: resin sealer

INTERVENTIONS:
Drug: bioceramic sealer — bioceramic based obturating sealer
  Other Names: endosequence
  Arms: endo sequence bioceramic sealer
Drug: MTA — MTA based obturating sealer
  Other Names: MTA fill apex
  Arms: MTA fill apex calcium silicate base sealer
Drug: resin sealer — resin based obturating sealer
  Other Names: AH Plus resin sealer
  Arms: AH plus resin sealer

SUMMARY:
aim of the study will be conducted to compare the effect of MTA fill apex sealer and endo sequence bioceramic sealer in obturation on the intenisty of postoperative pain and the incidence of post operative swelling in patient with necrotic teeth .

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring root canal treatment of single canal necrotic teeth.
* Patient from 18 to 60 years old
* Patients with Asymptomatic apical periodontitis.
* Teeth presenting with no clinical symptoms and with a periapical score from 2 to 4 according to Orstavik et al

Exclusion Criteria:

* Teeth with incompletely formed apex

  * Teeth requiring retreatment
  * Patients having complicating systemic disease such as diabetes, malignancy, pregnancy, central nervous system disorders, Cardiovascular system disorders, respiratory disorders, asthma patients, psychiatric disorders, immunocompromised patients
  * Patients taking anti-inflammatory or antibiotics
  * Patients giving history of analgesic or antibiotic intake 1 week before treatment
  * Patients below 18 years of age
* Patients above 65 years of age

  * Patients having history of peptic ulcer or gastrointestinal bleeding
  * Teeth affected with periodontal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-30 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Intensity of post-operative pain | 6 hours
  Measurement of post-operative pain by Visual analogue scale
Intensity of post-operative pain | 12 hours
  Measurement of post-operative pain by Visual analogue scale
Intensity of post-operative pain | 24 hours
  Measurement of post-operative pain by Visual analogue scale
Intensity of post-operative pain | 48 hours
  Measurement of post-operative pain by Visual analogue scale
Intensity of post-operative pain | 72 hours
  Measurement of post-operative pain by Visual analogue scale

SECONDARY OUTCOMES:
post operative swelling | 24 hours
  Yes or no yes or no